CLINICAL TRIAL: NCT05086718
Title: Composite Cartilage Perichondrium Graft for Air Bone Gap Closure in Chronic Suppurative Otitis Media Without Posterior Meatal Flap
Brief Title: Composite Cartilage Perichondrium Graft for Air Bone Gap Closure in Chronic Suppurative Otitis Media (CSOM) Without Posterior Meatal Flap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital Quetta (Other)
Responsible Party: Principal Investigator, Dr Zeeshan Ayub, Associate Professor ENT, Combined Military Hospital Quetta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRB/531/CMH Quetta
Record Dates: First submitted 2021-09-25; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Intervention Model Description: 300 cases of dry perforation CSOM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AB Gap Closure (Other): Air Bone gap closure following surgery will be considered as successful outcome
  Interventions: Other: Endoscopic ear surgery

INTERVENTIONS:
Other: Endoscopic ear surgery — Endoscopic approach without posterior meatal flap elevation will be employed in the ear with dry chronic suppurative otitis media. Tympanoplasty utilizing composite cartilage-fascia graft will be performed. After three months of time period successful outcome will be taken as closure of air bone gap on pure tone audiometry.

SUMMARY:
Composite Cartilage Perichondrium Graft for tympanoplasty in chronic suppurative otitis media (CSOM) Air Bone Gap (AB Gap) Closure will be taken as successful outcome Endoscopic technique without posterior meatal flap elevation

DETAILED DESCRIPTION:
300 eligible cases of dry CSOM will under go Composite Cartilage Perichondrium Graft tympanoplasty. Air Bone Gap Closure will be taken as successful outcome. The procedure will employ endoscopic technique without posterior meatal flap elevation.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders between 21 to 55 years
2. Dry chronic suppurative otitis media
3. Air bone gap between 15 to 25 Deci bel

Exclusion Criteria:

1. Discharging ear
2. Pediatric population
3. Ossicular Necrosis
4. Previous ear surgery

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Successful air bone gap closure on pure tone audiometry | Three months
  Three months of endoscopic tympanoplasty using composite cartilage-fascia graft, pure tone audiometry will be carried out measuring both air and bone conduction. Successful outcome will be closure of the air bone gap as compared with pre surgery air bone gap.

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Quetta, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
It will depend upon study outcome

REFERENCES:
- [Result] Akyigit A, Sakallioglu O, Karlidag T. Endoscopic tympanoplasty. J Otol. 2017 Jun;12(2):62-67. doi: 10.1016/j.joto.2017.04.004. Epub 2017 Apr 28. PMID 29937839